CLINICAL TRIAL: NCT05897047
Title: Prospective, Randomized Controlled Trial to Investigate Additional Interventional Telemedical Management Versus Standard Aftercare in Kidney Transplant Recipients (smartNTx)
Brief Title: The smartNTx Trial: A Prospective, Randomized Controlled Trial (RCT) to Investigate Additional Interventional Telemedical Management Versus Standard Aftercare in Kidney Transplant Recipients (KTR)
Acronym: smartNTx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01NVF21116; 0673 (Other: Universitätsklinikum Erlangen)
Record Dates: First submitted 2023-05-15; First posted 2023-06-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant Failure
Keywords: Aftercare; Telemedical Management

STUDY DESIGN:
Intervention Model Description: Prospective, two-armed randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group "Additional telemedical management" (Experimental): Patients in the interventional arm will receive a predefined additional telemedical management including regular telemedicine visits and automatic data transfer (e.g. vital signs, well-being, medication plan laboratory data and chat) between the patient at home and KTC through a certified smartphone application.
  Interventions: Combination Product: Additional interventional telemedical management
- Control group "Routine posttransplant aftercare" (No Intervention): Patients in the control group will receive routine posttransplant aftercare.

INTERVENTIONS:
Combination Product: Additional interventional telemedical management — Predefined additional telemedical management including regular telemedicine visits and automatic data transfer (e.g. vital signs, well-being, medication plan laboratory data and chat) between the patient at home and KTC through a certified smartphone application.
  Arms: Intervention group "Additional telemedical management"

SUMMARY:
The smartNTx trial: Prospective, randomized controlled trial (RCT) to investigate additional interventional telemedical management versus standard aftercare in kidney transplant recipients (KTR).

STUDY PURPOSE: To demonstrate that additional interventional telemedical management will lead to a higher chance for long-term graft survival, increase adherence, quality of life (QoL), and reduce complications and healthcare costs after kidney transplantation.

DETAILED DESCRIPTION:
This is a 1-year, prospective, randomized, 2-armed, parallel group multicenter trial in 3 German Kidney Transplant Centers (KTCs) to demonstrate that additional and continuous interventional telemedical management will lead to a better composite endpoint of 7 key outcome variables (hospitalizations, length of hospitalization, development of a de-novo donor specific antibody (DSA), medication adherence, tacrolimus intra-patient variability, blood pressure control and renal function after kidney transplantation). All patients will receive the same routine posttransplant aftercare. Patients in the interventional arm will receive a predefined additional telemedical management including regular telemedicine visits and automatic data transfer (e.g. vital signs, well-being, medication plan laboratory data and chat) between the patient at home and KTC through a certified smartphone application (comjoo business solutions GmbH, Berlin, Germany). Furthermore, home nephrologists of patients in the interventional arm are invited to participate in automatic data transfer of key variables (such as vital signs, laboratory data) with KTC. A separate telemedicine team will constantly review the incoming data according to a predefined protocol and eventually contact the patient and/or the home nephrologist in order to start appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation within last 12 months
* Treatment with tacrolimus
* Routine aftercare planned at KTC
* Ability to use a smartphone or tablet or with help of someone close by
* For children < 12 years parents have to take over the use of the smartphone
* Patients who are willing and able to participate in the study and from whom written informed consent has been obtained prior to study participation or pediatric patients with parenteral consent
* Ability to communicate in German or English
* Adequate and stable renal function (eGFR > 30 ml/min, Proteinuria < 1g/g creatinine) eGFR will be determined according to CKD-EPI for adults [81] or Schwartz formula for children [82]

Exclusion Criteria:

* Patient with mental dysfunction or inability to comply with the study protocol or pediatric patients whose parents cannot comply with the study protocol
* Any significant diseases or clinically significant findings, including psychiatric and behavioral problems, medical history and/or physical examination findings that would in the opinion of the investigator preclude the patient from participating in the study
* History of alcohol or drug abuse with less than 6 months of sobriety
* Participation in any other interventional clinical trial less than 1 month before participation in this study
* Patients who have been institutionalized by official or court order
* Patients with a combined kidney transplant or multi-organ recipients (other solid organ (e.g. pancreas) or bone marrow)
* Presence of DSA with MFI > 1000 at time of transplantation
* Recurrence of underlying kidney disease (e.g. focal segmental glomerulosclerosis (FSGS) or atypical hemolytic uremic syndrome (aHUS)
* Patient with active malignancy post-transplant with the exception of local, non-invasive, fully excised, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical carcinoma in situ
* Patients with clinically symptomatic congestive heart failure (CHF) or symptomatic coronary artery disease
* Patients with documented (either by serology and/or nuclear acid testing (NAT) clinically active infections (e.g. with a known hepatitis B (HBV), hepatitis C (HCV), HIV, CMV or BK virus infection).

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  According to BAASIS questionnaire at month 12
Unplanned hospitalizations | 12 months
  yes/no during study period
Length of unplanned hospitalization | 12 months
  More/less than 10 nights during study period
Development of de-novo DSA | 12 months
  yes/no at month 12
Tacrolimus intra-patient variability | 12 months
  Above/below 30% between month 6 to 12
Blood pressure control | 12 months
  normal/abnormal 24h-RR profile at month 12
Renal function | 12 months
  suboptimal renal function (eGFR < 45 ml/min at month 12

SECONDARY OUTCOMES:
Reduced graft losses (result evalution) | 12 months
  Documentation of graft losses at all visits - Month 3, 6, 9, 12
Better prognosis of the iBox score (result evalution) | 12 months
  Documentation of the prognosis of the AI during visit 5, month 12
Improvement in quality of life (result evalution) | 12 months
  Change in quality of life over 12 months (PROMIS 29 questionnaire) at month 0, 3, 6, 9, 12 (visit 1 to 5).
Improving disease management (process evalution) | 12 months
  Change in disease management over 12 months (PAM13 questionnaire) at month 0, 3, 6, 9, 12 (visit 1 to 5)
Acceptance of the new restoration among patients (process evalution) | 12 months
  Survey using established questionnaires and rating and satisfaction with care (own development) at Visit 4, 5 (month 9; 12)
Acceptance of the new restoration among service providers (process evalution) | 12 months
  Survey using established and newly developed questionnaires, as well as analyzes for usage behavior, including Grade and Assess Predictive tools. Benefit assessment of the data- and AI-supported Decision support (in-house development).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Schiffer, Prof. Dr., Principal Investigator — Uniklinikum Erlangen
Locations (2):
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin, Bavaria
  - University Hospital Essen, Essen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schiffer M, Pape L, Wolff JK, Gertges R, Visconti V, Reichert K, Pfau A, Dieterle A, Sauerstein K, Kribben A, Boss K, Karaterzi S, Nensa F, Winneckens P, Cypko M, Duettmann W, Zukunft B, Schrezenmeier E, Naik MG, Halleck F, Roller R, Moller S, Amft O, Budde K. The SmartNTx-study: a prospective, randomized controlled trial to investigate additional interventional telemedical management versus standard aftercare in kidney transplant recipients. Front Nephrol. 2025 Jun 19;5:1591962. doi: 10.3389/fneph.2025.1591962. eCollection 2025. PMID 40612527